CLINICAL TRIAL: NCT06794411
Title: Co-design, Implementation, and Evaluation of a Program to Promote Healthy Eating and Physical Activity Among Families in Situations of Social Vulnerability Linked to the Socio-educational Intervention Services of the Osona County Council.
Brief Title: Promotion of Healthy Eating Habits and Physical Activity Among Children and Their Families.
Acronym: ALIAFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: The Social Services Administration (Unknown)
Responsible Party: Principal Investigator, Cristina Vaqué, Principal Investigator, University of Vic - Central University of Catalonia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24/092
Record Dates: First submitted 2025-01-11; First posted 2025-01-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Families; Children; Food Habits; Physical Activity
Keywords: intervention; Family-based intervention; health promotion; children; Nutrition and physical activity; Social Vulnerability
MeSH Terms: conditions — Feeding Behavior; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pilot study with control group, not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Food habits and physical activity program.
  Interventions: Behavioral: Intervention group: Food habits and physical activity program
- Control group (Other): Usual care.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Intervention group: Food habits and physical activity program — 5 dynamic face-to-face sessions to promote healthy eating and regular physical activity. The 5 sessions are structured based on the pedagogical approach of Seeing, Judging and Acting (Gibson, 1999; Rodríguez-Bailón, et al., 2016). This methodology provides a logical structure to achieve nutritional and physical activity self-analysis. It is applied based on 3 stages:
  * 1st reflective stage: to raise awareness about the importance of following healthy eating and physical activity habits and identify to what extent families are close to the healthy recommendations in relation to these two habits (first two sessions).
  * 2nd: more active stage, to acquire strategies and learn to put these recommendations into practice in their day-to-day lives (session 3th and 4th session).
  * 3th: to plan specific actions to address and transform some aspects of improvement by freely assuming one's own commitment proposals with the aim of modifying the presented reality, if deemed appropriate (last session).
  Other Names: Nutrition and physical activity education
  Arms: Intervention group
Behavioral: Usual Care Group — They will be evaluated on baseline, final and follow up, and they will recieved basic nutritional and physical activity information.
  Arms: Control group

SUMMARY:
Eating habits and physical activity are key determinants of individual health. The family plays a relevant role in educating children about healthy lifestyles. In the Moroccan community, women are the reference for aspects related to family care. The main aim of this study is to evaluate the effect of the ALIAFF program on awareness and promotion of healthy eating and the practice of regular physical activity in families with a situation of social vulnerability linked to the socio-educational intervention services of the Osona County Council (CCO).

Children aged 9-12 years, along with their reference adult linked to the CCO's Socio-educational Intervention Services (SIS) with low adherence to the Mediterranean diet and/or low physical activity levels, with an interest to participate in the program who are able to independently reach the municipal centre.

The study involves participating in an initial meeting to co-create and culturally adapt the program. Following this, selected participants will complete the initial data collection with the help of a mediator of Moroccan origin. The intervention group will participate in five nutrition and physical activity sessions of 1.5 hours. After the intervention, both the control and the intervention group will participate in the final evaluation, which will also be repeated after two months to assess the longer-term impact. Upon completion of the evaluation, the control group will also receive the intervention as compensation for their participation.

DETAILED DESCRIPTION:
The intervention will start with the dissemination and recruitment phase. During this phase, the research team will provide detailed information about the project to the staff of Osona County Council (CCO) and Socio-educational Intervention Services (SIS). These staff members will then assist in identifying and inviting eligible children and one adult of their family (primarily mothers) who comply with the study's eligibility criteria. The municipal team will organize a meeting at SIS headquarters with the selected participants to facilitate extended information about the research and outline what their participation will entail. Families who agree to participate will be asked to sign the informed consent. This meeting will also serve as a collaborative space where families from both the control and the intervention groups can discuss the suitability of the proposed activities, session content, timetables, and interest dynamics of the families in order to co-create and culturally adapt the program. After that, the initial assessment will be conducted by the research team with the help of a mediator from the Moroccan community and the municipal social team through the initial data collection questionnaire (QRD). The intervention consisted of 5 dynamic face-to-face sessions of 1.5 hours will be implemented first with the intervention group. The sessions will be conducted by the researcher with the support of the social teams and a mediator of Morrocan origin in the SIS spaces of the municipality. The support material of every session will be provided to the participants and at the end of each session, small tasks will be assigned to encourage the transfer of the topics discussed during the sessions into the families' daily routines. The control group will receive the same intervention after the final evaluation as compensation for their participation in the program. At the end of the educational sessions, the final evaluation will be carried out for both groups through the final QRD. The same evaluation procedure will be repeated after two months to assess the program's impact and sustainability over time.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-12, along with their reference adult linked to the CCO's SIS (using the RUMI social diagnosis tool).
* Low adherence to the Mediterranean diet and/or low physical activity levels in either the child or the reference adult.

  * For children <3 points of KIDMED indicate a low level of adherence to the Mediterranean diet.
  * For adults <5 points of MEDAS indicate low adherence to the Mediterranean diet.
  * Through IPAQ fewer than three days of vigorous physical activity, five days of moderate physical activity, or walking less than 30 minutes per day are considered low physical activity levels.
* Having an interest in participating in a group program.
* Ability to independently reach the municipal centre.

Exclusion Criteria:

* Basic diagnosis of a serious intellectual developmental disorder that could make it impossible to follow the proposed sessions.
* Clinical contraindications for the practice of physical activity.
* Following a medically established dietary guideline that is incompatible with the Mediterranean diet.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Physical activity practice | Baseline (before study started), up to 5 weeks (through study completion)
  The International Questionnaire of Physical Activity - short version (IPAQ-SF) is the short version of the IPAQ (Craig et al., 2003), validated in Spain by Roman-Viñas et al. (2010).It measures, through 7 questions, the physical activity (vigorous, moderate and light) and the sitting time, and provide data for the total minutes of physical activity per week and the amount of sitting time per day.
Adults adherence to the Mediterranean diet | Baseline (before study started), up to 5 weeks (through study completion)
  Identified through a Mediterranean Diet Adherence Screener (MEDAS). Is a validated 14-item scale (Schröder et al., 2011) that assess questions related to food intake and frequency of consumption of foods that are typical and non-typical of the Mediterranean diet. The questions are dichotomous on habitual intakes of several food items. Responses that are favourable to the adoption of the Mediterranean diet score as 1 point, while response unfavourable are scored as 0. The final score ranges from 1 to 14. A score greater than 9 means high adherence to the Mediterranean diet.
Child adherence to the Mediterranean diet | Baseline (before study started), up to 5 weeks (through study completion)
  The KIDMED test (Mediterranean Diet Quality Index for children and teenagers) is a tool to evaluate the adherence to the mediterranean diet for children and youths.
  It was developed and validated by Serra-Majem et al. (2001). The index ranges from 0 to 12 and is based on a 16-questions test that can be self-administered or conducted by interview (pediatrician, dietitian, etc.). Questions denoting a negative connotation with respect to the MD are assigned a value of -1, and those with a positive aspect +1. The sums of the values from the administered test are classified into three levels: 1) >8, optimal Mediterranean Diet; 2) 4-7, improvement needed to adjust intake to Mediterranean patterns; 3) ≤3, very low diet quality.
Nutrition literacy | Baseline (before study started), up to 5 weeks (through study completion)
  2-item about nutritional knowledge measured by: true, false, I don't know, and 2 about nutritional skills measured with 5 points Likert scale were 1 is very easy and 5 is strongly difficult.
Physical activity literacy | Baseline (before study started), up to 5 weeks (through study completion)
  2-item about physical activity knowledge measured by: true, false, I don't know, and 2 about physical activity skills measured with 5 points Likert scale were 1 is very easy and 5 is strongly difficult.
Atitude towards healthy food habits and physical activity | Baseline (before study started) 5 weeks 8 weeks (through study completion)
  Lima-Serrano et al. (2012) questionnaire: 18 ítems. 5 point Likert scale where 1 is totally disagree and 5 is totally agree.

SECONDARY OUTCOMES:
Socio-demographic | Baseline
  Sex/Gender (female, male, non binary) Age (month and year of birth) Country of birth (name) Education status
Food allergies | Baseline
  No, yes.
Limitations to practice physical activity | Baseline
  No, yes
Health perception | Baseline (before study started), up to 5 weeks (through study completion)
  Visual analog scale, EuroQol (EQ-SD) were 0 means the worst health you can imagine, and 100 the best health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina V Vaque Crusellas, Doctrate, Principal Investigator — University of Vic-University Central of Catalonia
Locations (1):
- Social Services of the Regional Council of Osona, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided